CLINICAL TRIAL: NCT06621927
Title: Effect of Ideal Food Pyramid on Gut Microbiota, Disease Activity, Body Composition and Biochemical Parameters in Rheumatoid Arthritis: A Randomized Controlled Trial
Brief Title: The Effect of the Ideal Food Pyramid on Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Betül Cicek, Prof.Dr., TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EU-BVD-UKM-02
Record Dates: First submitted 2024-09-18; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Gut Microbiota; Ideal food pyramid; rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Diet

STUDY DESIGN:
Intervention Model Description: two separate groups simultaneously diet and control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group receiving nutritional intervention (Active Comparator): The ideal food pyramid created for rheumatoid arthritis patients was applied to the patients and followed for 12 weeks.
  Interventions: Other: Diet
- control group (Placebo Comparator): Patients diagnosed with rheumatoid arthritis and meeting the inclusion criteria were included in the control group and no intervention was applied. At the beginning and end of the study, a questionnaire, blood and stool samples were taken.
  Interventions: Other: Control (Standard treatment)

INTERVENTIONS:
Other: Diet — The Ideal Food Pyramid, which has not been applied before, is used to observe disease activities and especially changes in intestinal microbiota in rheumatoid arthritis.
  Arms: Group receiving nutritional intervention
Other: Control (Standard treatment) — We chose a control group to show the effect of the intervention we would apply to the diet group and did not apply any intervention to the control group.
  Arms: control group

SUMMARY:
The aim of this study was to observe the effects of the Ideal Food Pyramid created for Rheumatoid Arthritis patients on disease activity, inflammatory markers, body composition and intestinal microbiota. The main questions it aims to answer are:

* Does the Ideal Food Pyramid improve dysbiosis in patients with rheumatoid arthritis?
* Does the Ideal Food Pyramid improve clinical and laboratory findings in patients with rheumatoid arthritis? Researchers will compare the Ideal Food Pyramid with a control group (no intervention) to determine if it has an effect on rheumatoid arthritis.

Participants:

All participants will fill out questionnaires at the beginning of the study, blood and stool will be collected. These procedures will be repeated at the end of the study.

Diet or control (no intervention) will be applied for 12 weeks Diet group will be checked for compliance with the diet every 2 weeks

DETAILED DESCRIPTION:
This study will be conducted on patients diagnosed with Rheumatoid Arthritis who meet the inclusion criteria and apply to the Rheumatology Polyclinic of Erciyes University Faculty of Medicine Hospital. Diagnosed patients will be directed to the Diet Polyclinic. Patients who come to the polyclinic will be included in the study on a voluntary basis and the patients will sign an informed consent form. A diet program based on the pyramid created for Rheumatoid arthritis patients will be created for each patient and will be followed for 12 weeks. A questionnaire form containing questions about sociodemographic characteristics, nutritional habits, anthropometric measurements, physical activity status and disease activity will be filled out by face-to-face interviews with the patients. The questionnaire and scale forms used for disease activity and physical activity status are as follows: DAS28 (Disease Activity Score), Simple Disease Activity Index (SDAI), Health Assessment Questionnaire (HAQ), International Physical Activity Questionnaire (Short), Visual Analog Scale (VAS), SF-36 Quality of Life Scale (Short Form 36), Rheumatoid Arthritis Quality of Life Scale (QOL-RA). Fecal samples, blood samples and anthropometric measurements will be taken from the volunteers before starting the study and twice at the end of 12 weeks, and comparisons will be made before and after. Fecal samples taken from individuals will be stored at -80°C until the day of analysis for microbiota analysis. The samples will be processed in the Metagenome laboratory at Erciyes University Genome and Stem Cell Center (GENKÖK) and sequenced using the 16s rRNA next generation sequencing method. The obtained data will be analyzed in detail with an artificial intelligence algorithm and reported. Blood will be taken from individuals after 10-12 hours of fasting; Fasting blood glucose (mg/dl), C reactive protein (CRP), sedimentation rate (mm/s), triglyceride (mg/dl), cholesterol (mg/dl), HDL cholesterol (mg/dl), LDL cholesterol (mg/dl), urea (mg/dl), creatinine (mg/dl), uric acid (mg/dl), complete blood count (hemogram), aspartate aminotransferase (AST) (IU/L), alanine aminotransferase (ALT) (IU/L) values will be checked at Erciyes University Central Laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria,

  1. Diagnosed with Rheumatoid Arthritis by a rheumatologist and starting disease-modifying antirheumatic drug (DMARD) treatment.
  2. Those with rheumatoid arthritis disease duration longer than 1 year
  3. Being between the ages of 18-65
  4. Body Mass Index (BMI)=18.5-40 kg/m2
  5. Smoking three or less cigarettes per day

Exclusion Criteria:

* Exclusion criteria

  1. Those with cancer, diabetes, kidney, inflammatory bowel disease, and liver disease, psychiatric disorders
  2. Those who use regular Non-Steroidal Anti-Inflammatory Drugs (NSAIDs), those whose oral cortisol intake is >12.5 mg
  3. Those who have used a special diet, herbal supplements, vitamin-mineral supplements (except for vitamin D), and probiotics in the last 3 months
  4. Those who have received antibiotic treatment in the last 3 months
  5. Those who are breastfeeding or pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Gut Microbiota | 12 week
  Pre- and post-study stool samples were collected from all participants. To ensure sample integrity, all collected samples were immediately stored at -80°C until further processing.
  The stages of microbiota analysis are listed below, respectively.
  1. DNA isolation from stool samples:
     - DNA extraction from stool samples was performed using the Qiagen Power Soil DNA Extraction Kit (Qiagen, Hilden, Germany). Quantification of double-stranded DNA (dsDNA) was performed using the Qubit dsDNA HS Assay Kit and a Qubit 2.0 Fluorimeter (Thermo Fisher Scientific, Waltham, MA, USA).
  2. Illumina miSeq 16S rRNA next-generation sequencing. Analysis features:
     * V4 variable region PCR amplification
     * Paired-end sequencing of 2 x 250 bp amplicons.
     * At least 50,000 reads per sample (>Q30 quality) Data on microbiota are given in order of taxonomic classification from phylum to genus level.

SECONDARY OUTCOMES:
C reactive protein (CRP) (mg/dL) | 12 week
  CRP was measured twice, at the beginning and at the end of the study, using the immunoturbidimetric method on the Cobos c701 (Roche Diagnostic- Basel, Switzerland) autoanalyzer.
Erythrocyte sedimentation rate (ESR) (mg/dL) | 12 week
  Sedimentation rate will be studied twice, at the beginning and at the end of the study, using a Vision C ESR autoanalyzer (Shenzhen, China).
Total cholesterol,(mg/dL) | 12 week
  Total cholesterol will be measured spectrophotometrically on a Cobos c701 (Roche Diagnostic-Basel, Switzerland) autoanalyzer at the beginning of the study and at the end of 12 weeks.
LDL cholesterol (mg/dL) | 12 week
  LDL cholesterol will be measured spectrophotometrically on a Cobos c701 (Roche Diagnostic-Basel, Switzerland) autoanalyzer at the beginning of the study and at the end of 12 weeks.
DAS28ESR | 12 week
  DAS28-ESR includes the number of tender and swollen joints in 28 joints, the patient's estimate of their general health on the VAS, and the ESR.
  • DAS28-ESR was calculated as 0.56 × √(Tender joint count) + 0.28 × √(Swollen joint count) + 0.7 × ln ESR + 0.014 × VAS-GH.
  The score ranges from 0 to 9.4; values exceeding 5.1 are indicative of active disease and scores <3.2 indicate an inactive, well-controlled disease state.
DAS28CRP | 12 week
  DAS28-CRP includes the number of tender and swollen joints in 28 joints, the patient's estimate of their general health on the VAS, and the CRP.
  • DAS28-CRP was calculated as 0.56 × √(Tender joint count) + 0.28 × √(Swollen joint count) + 0.36 × ln (CRP + 1) + 0.014 × VAS-GH + 0.96 The score ranges from 0 to 9.4; values exceeding 5.1 are indicative of active disease and scores <3.2 indicate an inactive, well-controlled disease state.
The Simple Disease Activity Index (SDAI) | 12 week
  SDAI is calculated as the numerical sum of tender and swollen joint patient global assessment, physician global assessment, and C-reactive protein (CRP) level (mg/dL), with scores ranging from 0 to 86; A score of ≤ 3.3 is defined as remission, >3.3 to ≤ 11 indicates low disease activity, >11 and ≤ 26 indicates moderate disease activity, and high disease activity is defined by scores >40.
The Health Assessment Questionnaire (HAQ) | 12 week
  HAQ consists of 20 questions in 8 categories. Questions are scored from 0 to 3, with higher scores indicating worse functioning. Joint pain was measured using a horizontal visual analog scale (VAS) ranging from 0 to 10; higher scores indicate greater pain.
The Rheumatoid Arthritis Quality of Life instrument (RAQoL) | 12 week
  RAQoL consists of 30 questions, and participants are asked to indicate whether each question applies to them. Scores range from 0 to 30, with higher scores indicating lower quality of life.
The 36-item Short Form Health Survey (SF-36) | 12 week
  SF-36 measures health-related quality of life using eight items: physical function, physical role difficulty, pain, general health perception, energy/vitality, social functioning, emotional role difficulty, and mental health. The SF-36 scales range from 0 to 100, with higher scores indicating better quality of life.
Body fat percentage | 12 week
  Body fat percentage is shown as a percentage (%). Measurement was made at the beginning and end of the study using a Tanita BC 418MA brand (bioelectrical impedance device [BIA]). For BIA measurement, individuals were asked not to do any heavy physical activity 24-48 hours before, not to consume alcohol 24 hours before, to come with at least 4 hours of fasting, not to consume too much liquid (water, tea, coffee) before the analysis (at least 4 hours) and not to carry any metal objects on them.
Body fat mass | 12 week
  Body fat mass is calculated in kilograms. Measurement was made at the beginning and end of the study using a Tanita BC 418MA brand (bioelectrical impedance device [BIA]). For BIA measurement, individuals were asked not to do any heavy physical activity 24-48 hours before, not to consume alcohol 24 hours before, to come with at least 4 hours of fasting, not to consume too much liquid (water, tea, coffee) before the analysis (at least 4 hours) and not to carry any metal objects on them.
Body mass index (BMI) | 12 week
  The formula "BMI=Weight (kg)/Height (m²)" was calculated.
Waist circumference (cm) | 12 week
  The person to be measured is standing on their right side and the lowest rib bone is found and marked. The hip bone protrusion (cristailiac) is found on the hip and marked. The circumference passing through the middle of the two marked points is measured with a non-stretchable tape measure.
Hip circumference(cm) | 12 week
  Hip circumference is measured with a non-stretchable tape measure at the widest part of the hip when viewed from the side while the individual is standing. It is written in centimeters.
Neck circumference (cm) | 12 week
  Neck circumference is measured with a tape measure passing from the point where the neck and shoulders meet, just below the larynx.
Wrist circumference (cm) | 12 week
  Wrist circumference is measured with subjects in a seated position using a tension-gated tape measure placed over Lister's tubercle of the distal radius and the distal ulna.
Hand grip strength (kg) | 12 week
  The Jamar hand dynamometer, recommended by the American Association of Hand Therapists (AETD) and accepted as the gold standard for many studies with high validity and reliability, was used to measure hand grip strength. During the test, they were informed not to hold their breath and not to shake the dynamometer. In order to determine the dominant hand, participants were asked which hand they used while eating or writing. Each hand was measured 3 times and the average was taken, with the patients in a sitting position, shoulder adduction and neutral rotation, elbow 90 degrees flexed, forearm in midrotation and supported wrist in neutral.

CONTACTS AND LOCATIONS:
Overall Officials: Ülger Kaçar Mutlutürk, Principal Investigator — Erciyes University Medical Faculty Hospital
Locations (1):
- Erciyes University Medical Faculty Hospital, Kayseri, Melikgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No